CLINICAL TRIAL: NCT03825146
Title: A Phase I Single-arm, Open-label Prospective Study to Evaluate the Efficacy and Safety of Peripheral Blood Derived Autologous Multi-lineage Potential Cells (AMPC) in Relapsed/Refractory Acute Myeloid Leukemia (AMPCAL Study)
Brief Title: The Effects of AMPC in the Treatments of Refractory or Relapsed AML
Acronym: AMPCAL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lai Corporation Pty. Ltd. (Industry)
Responsible Party: Principal Investigator, Supachai Ekwattanakit, Principle Investigator, Lai Corporation Pty. Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOP-PNC-REC-01/01-061
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Acute Myeloid Leukaemia Recurrent
Keywords: relapse/refractory acute myeloid leukaemia; autologous progenitor cells
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Single-arm, open label, prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (AMPC) (Experimental): AMPC will be intravenously infused.
  Interventions: Biological: Autologous Multi-lineage Potential Cells (AMPC)

INTERVENTIONS:
Biological: Autologous Multi-lineage Potential Cells (AMPC) — Multi-lineage potential cells which were induced to de-differentiate from somatic leukocytes from peripheral blood. Cells are autologous with respect to the patient, and are prepared in a suspension and administered via intravenous infusion.
  An estimated average of 1 x 10^8 (0.5 to 5.0 x 10^8) cells/per suspension(275 to 450mL) will be infused into the patient via intravenous infusion on day 5. Cell counts depend on yield of initial leukocyte harvest on day 0.

SUMMARY:
A private trial for evaluating the overall response rate contributed by AMPC in AML in refractory or relapsed AML

DETAILED DESCRIPTION:
After inclusion and exclusion criteria has been determined and approved, written informed consent will be obtained from the candidate. All medical history relevant to the diagnosis of AML will be collected.

Screening period:

The screening period could extend from 0 to 7 days depending on the completion of screening laboratory results as below.

On day -5 (up to day -1), the patient will undergo a screening test for the following test items:

* BUN, creatinine, electrolyte, liver function test (LFT)
* Full blood count (FBC), including blood smear
* Hepatitis B/C
* Human T lymphocytic virus type I and II (HTLV-I/II)
* HIV1/2
* Syphilis serology
* Mycoplasma serology For Hepatitis B/C,HTLV-I/II, HIV1/2, Syphilis serology, and Mycoplasma serology, these tests obtained up to 3 months prior to day -5 can be allowed for using as screening result.
* Chest X-ray
* Bone marrow study including aspiration with wright's stain, biopsy, flow cytometry, and chromosome study (Any molecular testing for AML is optional.).

Bone marrow biopsy can be omitted if the prior study performed within 14 days before day-5 and the available materials (core biopsy and slides) and result can be obtained for pathological review. In this case, only bone marrow aspiration for Wright's stain, flow cytometry, and chromosome study will be performed.

Bone marrow biopsy will be repeated if the previous result has been performed more than 14 days prior to day -5 and/or FBC at day -5 reveals peripheral blast count higher than 10% of total white blood cells.

For chromosome study (cytogenetics), the previous result before the recent line of chemotherapy prior to enrollment can be used for the screening data.

On day 0, peripheral blood will then be collected, ranging from 250mL to 400mL depending on candidate fitness. The blood is collected into a sterile blood bag and sealed. Subsequent processes will be conducted in the blood bag within a closed-system to minimize contamination risks. FBC will be collected in order to determine the disease status. After that, the investigator will consider to prescribe blood transfusion for the candidate.

On day 0 to day 3, the collected blood will be sent to the laboratory for stem cell culture, and a sample of the collected blood will be sent to a third-party laboratory for contamination testing of the following parameters:

* Bacterial endotoxin
* Total viable aerobic count
* Total viable count
* Microbial growth
* Mycoplasma real-time PCR test

On day 4, the biotest results will be released and the safety profiles of the AMPC product must be completed and passed before the cultured stem cells may be released for treatment

On day 5, candidates will receive an infusion of the cultured stem cells. Prior to the infusion, FBC and blood chemistry (BUN, Cr, electrolyte, LFT) will be collected and the treating doctor will first conduct an allergy skin test to determine suitability for reinfusion. The cultured stem cells are then reinfused intravenously into the candidate in a process that could take up to 2 hours

The candidate participation will take place on day 0 to day 1 or 2 (if blood transfusion is required) and day 5 (period adjusted for blood transfusion if required) for peripheral blood collection and stem cell reinfusion respectively; with 12 month follow up after treatment;

* 3 days post-treatment follow-up: full blood count test and blood smear, BUN, Cr, electrolyte, LFT
* 10 days post-treatment follow-up: full blood count test and blood smear, BUN, Cr, electrolyte, LFT
* 1 month (+/-7 days) post-treatment follow-up: full blood count test and blood smear, BUN, Cr, electrolyte, LFT, bone marrow study
* 3 month (+/-7 days) post-treatment follow-up: full blood count test and blood smear, BUN, Cr, electrolyte, LFT, bone marrow study
* 6 month (+/-7 days) post-treatment follow-up: full blood count test with bone marrow study
* 12 month (+/-7 days) post-treatment follow-up: full blood count test with bone marrow study

ELIGIBILITY:
Inclusion Criteria:

* Must be unequivocally diagnosed with AML according to WHO classification with accompanying bone marrow biopsy and blood panel results
* Must have refractory AML, defined as disease unresponsive to initial treatment; or relapsed AML that re-occured after treatment with conventional high dose chemotherapy
* Candidates who have no available match-sibling donor for bone marrow transplantation (BMT) or are not suitable for BMT due to any reason.
* Must have had prior treatment with chemotherapy at least 30 days prior to day 0 of this study and have recovered from treatment-related toxicity of chemotherapeutic agents with the exception of persistent diseases
* Age 20 to 60 years old

Exclusion Criteria:

* Candidates who received any investigational therapies 4 weeks prior to treatment with this protocol
* Candidates who received radiotherapy within 4 weeks prior to the treatment of this protocol
* Candidates who have not recovered from any AE caused by radiotherapy or any agents received 4 weeks earlier
* Candidates who have had a prior allogeneic stem cell transplant
* Known case of extramedullary myeloid tumor (myeloid sarcoma)
* Pregnant or breastfeeding women
* Hydroxyurea has been prescribed within 10 days prior to day-5
* Candidates have any abnormal screening laboratory results as below;

  * Hemoglobin < 9 g/dL
  * Total white blood cells count > 30,000/microL (without ongoing G-CSF therapy)
  * Platelet count < 75,000/microL
  * Creatinine clearance < 30 mL/min/1.73 m2 (by Cockcroft and Gault formula)
  * ALT > 5x upper normal limit
  * Bone marrow study at screening period show blast > 40% of total nucleated cells or severe hypocellularity (defined as < 25% of normal cellularity for corresponding age) with presence of cluster of blasts
* Candidates have active heart disease including recent or chronic heart failure, unstable angina, recent acute myocardial infarction, or significant arrhythmia within 6 months of recruitment.
* Candidates have concurrent malignancies unless the candidates has been free of the disease for at least 5 years.
* Candidates positive for HIV1/2, hepatitis B/C, HTLVI/II, and Syphilis

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-01-04 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) of AMPC in refractory/relapsed AML at 12 months | 12 months
  Overall response rate (ORR) is defined as whether the patient achieves complete remission (CR) or complete remission with incomplete blood count recovery (CRi)
  CR Requirements:
  * Bone marrow aspiration shows less than 5% of abnormal blasts as determined by evidence from flow cytometry or immunohistochemistry
  * Bone marrow biopsy shows no clusters of blast cell
  * Normal values for absolute neutrophil count in peripheral blood exceeds 1,000/microL
  * Platelet count in peripheral blood exceeds 100,000/microL
  * Absence of extramedullary AML
  CRi Requirements:
  * All parameters of CR except platelet recovery or neutrophil recovery
  * Incomplete recovery-platelet count is less than 100,000/microL or neutrophil count less than 1,000/microL in peripheral blood

SECONDARY OUTCOMES:
Safety profile and treatment-related adverse events (AE) upto 12-month follow up period | 12 months
  AE is defined as any unintended or undesirable experience that occur during the course of the clinical investigation regardless of whether they are considered to be drug-related.
ORR of AMPC in refractory/relapsed AML at 3 and 6 months | 3 and 6 months
Overall survival (OS) rate at 12 months | 12 months
Time-to-next treatment (TTNT), defined as the time from the start of AMPC therapy to the start date of a subsequent line of therapy. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Supachai Ekwattanakit, Ph.D, M.D., Principal Investigator — Panacee Hospital Rama 2
Locations (1):
- Panacee Hospital Rama 2, Samut Sakhon, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT03825146/Prot_SAP_000.pdf